CLINICAL TRIAL: NCT04789616
Title: The CAMAROS Trial: The Canadian Maraviroc Randomized Controlled Trial To Augment Rehabilitation Outcomes After Stroke
Brief Title: The Canadian Maraviroc Randomized Controlled Trial To Augment Rehabilitation Outcomes After Stroke
Acronym: CAMAROS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University Health Network, Toronto (Other); University of California, Los Angeles (Other); Sunnybrook Health Sciences Centre (Other); University of British Columbia (Other); Memorial University of Newfoundland (Other); Dalhousie University (Other); Parkwood Hospital, London, Ontario (Other); Riverview Health Centre Foundation (Other); The Dr. Miriam and Sheldon G. Adelson Medical Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB21-0258
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Rehabilitation; Exercise; Maraviroc; Randomized Control Trial; Activity Sensors; Motor Learning; Retention; Wearable Sensors; Celsentri
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Maraviroc; Resistance Training; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maraviroc (Celsentri) (Experimental): Maraviroc (Celsentri) will be administered to this group. Participants will be administered a dose of 300mg to be taken twice per day for the duration of the exercise intervention (8 weeks).
  Interventions: Drug: Maraviroc; Behavioral: Exercise Program; Device: Activity Sensor; Behavioral: Motor Learning
- Placebo (Placebo Comparator): An over-encapsulated placebo, or "sugar pill" (so it appears identical to the trial drug) will be administered to this group. Participants will be administered the placebo identical to the 300mg maraviroc tablet for the duration of the exercise intervention (8 weeks).
  Interventions: Behavioral: Exercise Program; Other: Placebo; Device: Activity Sensor; Behavioral: Motor Learning

INTERVENTIONS:
Drug: Maraviroc — Half of the participants will take maraviroc for a period of 8 weeks.
  Other Names: Celsentri
  Arms: Maraviroc (Celsentri)
Behavioral: Exercise Program — All participants will take part in an 8-week exercise program. While in-hospital, participants will undergo standard of care rehabilitation (estimated at 45 minutes each daily for physiotherapy & occupational therapy) plus a supplementary upper extremity exercise program (Graded Repetitive Arm Supplementary Program (GRASP); estimated at 1 hour daily).
  After discharge from inpatient care, participants will complete an at-home supplementary upper and lower extremity exercise program. This program will include 30 minutes daily walking or sit-to-stand exercises and 30 minutes daily practice using the GRASP program.
Other: Placebo — Half of the participants will take a placebo for a period of 8 weeks.
  Other Names: "Sugar" Pill
  Arms: Placebo
Device: Activity Sensor — Participants will be asked to wear small activity sensors (one on each wrist and one on each ankle, total of four sensors) at the baseline, 4-week, 8-week, and 6-month assessments for 7 consecutive days. Activity related to walking, sleep, physical activity, and arm and leg movement throughout the day will be measured.
  The sensors will be worn for a total of 28 days throughout the study.
Behavioral: Motor Learning — Participants will be asked to perform a computer-based motor learning assessment at the baseline, 4-week, 8-week, and 6-month assessments. A retention task, which involves shorter versions of the initial tasks, will also be completed within 72 hours of the initial assessment (initial test and retention test).

SUMMARY:
The CAMAROS trial is a randomized controlled phase II trial analyzing the effect of coupling a C-C chemokine receptor 5 (CCR5) antagonist, Maraviroc (Celsentri), and exercise to improve both upper and lower extremity recovery after a stroke.

DETAILED DESCRIPTION:
After stroke, the combination of progressive skills practice in an adequate dose plus exercise for fitness augments motor and cognitive outcomes. However, sensorimotor and cognitive improvements often plateau after 12 weeks. There is an urgent need to find novel methods to drive recovery and lessen limb paralysis. Drugs that might enhance learning or neural repair, as well as other molecular and synaptic adaptations that occur during skills training and fitness exercise, might extend that recovery curve, although to date only fluoxetine has given any hint of this. Most trials have tested agents that modulate neurotransmitters. Several very recent preclinical experiments and observational studies in patients after stroke suggest that the commercially available medication, Maraviroc, may augment skills learning during rehabilitation training especially during the first three months after onset, by acting on unique molecular components for novel learning.

The CAMAROS trial is a randomized, placebo-controlled, blinded phase II trial evaluating the efficacy of coupling Maraviroc (Celsentri) with exercise rehabilitation across multiple Canadian sites in 120 stroke participants. Patients will begin their participation within 8 weeks of stroke onset. Both groups will receive an exercise program in addition to standard of care rehabilitation, but only one group (the intervention group) will receive the active drug Maraviroc.

Study participants will be evaluated using physical assessments, cognitive assessments, and using wrist and ankle activity sensors at baseline, after 4 weeks of taking the drug/placebo, after 8 weeks of taking the drug/placebo, and at 6-months post-stroke. While enrolled in the study, participants will be required to take part in an 8 week, daily exercise program. Participants will also perform a short motor learning assessment at each formal assessment and again within 72 hours of each formal assessment (initial test and retention test).

Evaluators and participants will be blind to the treatment administered. The trial is constructed with randomization to remove selection and allocation biases and to ensure greater validity in observed differences in the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Primary ischemic anterior circulation stroke
2. Age ≥18 years
3. At least 5 days after stroke but within 8 weeks of stroke on the date of medication (maraviroc or placebo) start
4. Hemiparesis requiring inpatient rehabilitation
5. Assistance available for daily rehabilitation training practice and for transportation when needed
6. Adequate language skills to understand the Informed Consent and retain information during daily therapies
7. At least one of the following:

   * some shoulder abduction with gravity eliminated and visible extension in two or more digits OR
   * visible hip flexion or extension

Subgroup Stratification Criteria

1. For Upper Extremity Group:

   * Minimum Ability: Medical Research Council (MRC) grade >1 for shoulder abduction AND MRC grade >1 for finger extensor on at least two digits
   * Maximum Ability: Upper Extremity Fugl-Meyer Assessment Score >56
2. For Lower Extremity Group:

   * Minimum Ability: requiring a 2-person assist
   * Maximum Ability: walking speed <0.8m/s

Exclusion Criteria:

1. Pre-stroke modified Rankin score ≥ 2
2. Limited resources or illness that will not enable a return to living outside of a facility
3. History of dementia
4. History of hepatitis or elevated hepatic transaminases or bilirubin
5. History of renal insufficiency or creatinine clearance (eGFR) < 60mL / min / 1.73m2
6. Cancer or other chronic illness that makes 1-year survival unlikely or will detract from the ability to carry out exercise and skills practice
7. Existing pre-stroke serious disabling disease (e.g., Parkinson's disease, severe traumatic brain injury, amputation)
8. Seizure related to stroke
9. Acute or chronic epilepsy
10. Currently taking any of the following anticonvulsant medications:

    * Carbamazepine
    * Phenobarbital
    * Phenytoin
11. Pregnant, breastfeeding, or positive test for pregnancy at baseline
12. Women of childbearing potential who are not using one highly effective form of contraception or two forms of effective contraception
13. Known HIV positivity
14. Currently taking any of the following antifungal and/or antibacterial medications:

    * Ketoconazole
    * Itraconazole
    * Voriconazole
    * Rifampin
    * Clarithromycin
    * Rifabutin + Protease Inhibitor
15. Currently taking St. John's Wort
16. Currently taking Paxlovid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Upper Extremity Assessment Score | Baseline (between 5 days and 8 weeks after stroke), after 4 weeks on drug/placebo, after 8 weeks on drug/placebo, and 6-months post-stroke
  Difference in subscale scores on the Upper-Extremity Fugl-Meyer Assessment - both motor (max 66) and sensory (max 12) components. Higher scores indicate better outcome.
Change in 10-Meter Walk Test Score | Baseline (between 5 days and 8 weeks after stroke), after 4 weeks on drug/placebo, after 8 weeks on drug/placebo, and 6-months post-stroke
  A performance measure used to assess walking speed in meters per second over a short distance. It can be used to determine functional mobility, gait, and vestibular function. Faster speed indicates better function.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline (between 5 days and 8 weeks after stroke), after 4 weeks on drug/placebo, after 8 weeks on drug/placebo, and 6-months post-stroke
  The ARAT assesses arm function to determine the quality of the arm movement, and the limitation of activity. The ARAT consists of 4 sub-tests; that examines and individual's grip, grasp, pinch and gross motor movement in order to determine upper extremity function. Objects of varying size, shape, and weight must be either grasped, handled or moved in a specific task in order to evaluate function. Low scores mean worse function with the minimum possible score being 0 and the highest possible score being 57 (normal function).
6 Minute Walk Test | Baseline (between 5 days and 8 weeks after stroke), after 4 weeks on drug/placebo, after 8 weeks on drug/placebo, and 6-months post-stroke
  An assessment of ambulatory function by measuring the distance walked over a period of 6 minutes. Greater distance walked indicates better function.

OTHER OUTCOMES:
Fugl-Meyer Lower Extremity Assessment Score | Baseline (between 5 days and 8 weeks after stroke), after 4 weeks on drug/placebo, after 8 weeks on drug/placebo, and 6-months post-stroke
  Fugl-Meyer Lower Extremity Assessment assesses motor and sensorimotor impairment in the lower extremities. Total score is between 0 and 34. Sub-scales include: proximal (0-18), knee/ankle (0-10) and coordination/speed (0-6). Higher scores indicate better performance. Sub-scale scores are summed to calculate total score.
Patient Health Questionnaire 9 (PHQ-9) | Baseline (between 5 days and 8 weeks after stroke), after 8 weeks on drug/placebo, and 6-months post-stroke
  A 9-question measurement used to screen for the presence and severity of depression.
Stroke Aphasia Depression Questionnaire (SADQ) | BaselineBaseline (between 5 days and 8 weeks after stroke), after 8 weeks on drug/placebo, and 6-months post-stroke, 8-week assessment, and 6-month assessment
  A 10-item questionnaire completed by a caregiver to quickly assess depressive symptoms in stroke patients with aphasia. Higher scores indicate a greater likelihood of depression.
European Quality of Life Across 5 Domains (EQ-5D) | Baseline (between 5 days and 8 weeks after stroke), after 8 weeks on drug/placebo, and 6-months post-stroke
  A self-completion questionnaire used to assess health-related quality of life.
Stroke Impact Scale (SIS) | Baseline (between 5 days and 8 weeks after stroke), after 8 weeks on drug/placebo, and 6-months post-stroke
  Stroke-specific, self-report, health status measure. Assesses multiple domains on a 5-point Likert scale. Domains include: strength (4-20), hand function (5-25), activities of daily living/instrumental activities of daily living (10-50), mobility (9-45), communication (7-35), emotion (9-45), memory and thinking (7-35), and participation (8-40). An extra question asks that the patient rate on a scale from 0 - 100 how much they feel that he/she has recovered from his/her stroke. The 4 physical domains (strength, hand function, mobility and activities of daily living) can be summed together to create a single, physical dimension score (28-140) while all other domains should remain separate. Higher scores indicate better function.
National Institutes of Health Stroke Scale (NIHSS) | Baseline (between 5 days and 8 weeks after stroke) and 6-months post-stroke
  A 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Higher scores indicate greater impairment.
Montreal Cognitive Assessment (MoCA) | Baseline (between 5 days and 8 weeks after stroke) and 6-months post-stroke
  A cognitive screening test used to assess: short term memory, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place. Higher scores indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Dukelow, MD PhD FRCPC, Principal Investigator — University of Calgary, Calgary, Alberta, Canada; Bruce Dobkin, MD, Study Chair — University of California, Los Angeles, California, USA
Locations (6):
- Canada (6):
  - University of Calgary & Foothills Medical Centre, Calgary, Alberta
  - University of British Columbia & GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Parkwood Institute, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben Assayag E, Korczyn AD, Giladi N, Goldbourt U, Berliner AS, Shenhar-Tsarfaty S, Kliper E, Hallevi H, Shopin L, Hendler T, Baashat DB, Aizenstein O, Soreq H, Katz N, Solomon Z, Mike A, Usher S, Hausdorff JM, Auriel E, Shapira I, Bornstein NM. Predictors for poststroke outcomes: the Tel Aviv Brain Acute Stroke Cohort (TABASCO) study protocol. Int J Stroke. 2012 Jun;7(4):341-7. doi: 10.1111/j.1747-4949.2011.00652.x. Epub 2011 Nov 2. PMID 22044517
- [Background] Ben Assayag E, Shenhar-Tsarfaty S, Korczyn AD, Kliper E, Hallevi H, Shopin L, Auriel E, Giladi N, Mike A, Halevy A, Weiss A, Mirelman A, Bornstein NM, Hausdorff JM. Gait measures as predictors of poststroke cognitive function: evidence from the TABASCO study. Stroke. 2015 Apr;46(4):1077-83. doi: 10.1161/STROKEAHA.114.007346. Epub 2015 Feb 12. PMID 25677599
- [Background] Ben Assayag E, Tene O, Korczyn AD, Shopin L, Auriel E, Molad J, Hallevi H, Kirschbaum C, Bornstein NM, Shenhar-Tsarfaty S, Kliper E, Stalder T. High hair cortisol concentrations predict worse cognitive outcome after stroke: Results from the TABASCO prospective cohort study. Psychoneuroendocrinology. 2017 Aug;82:133-139. doi: 10.1016/j.psyneuen.2017.05.013. Epub 2017 May 18. PMID 28549269
- [Background] Dobkin BH. A Rehabilitation-Internet-of-Things in the Home to Augment Motor Skills and Exercise Training. Neurorehabil Neural Repair. 2017 Mar;31(3):217-227. doi: 10.1177/1545968316680490. Epub 2016 Nov 24. PMID 27885161
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK, Cen S, Hayden SK; LEAPS Investigative Team. Body-weight-supported treadmill rehabilitation after stroke. N Engl J Med. 2011 May 26;364(21):2026-36. doi: 10.1056/NEJMoa1010790. PMID 21612471
- [Background] Hiragami S, Inoue Y, Harada K. Minimal clinically important difference for the Fugl-Meyer assessment of the upper extremity in convalescent stroke patients with moderate to severe hemiparesis. J Phys Ther Sci. 2019 Nov;31(11):917-921. doi: 10.1589/jpts.31.917. Epub 2019 Nov 26. PMID 31871377
- [Background] Joy MT, Ben Assayag E, Shabashov-Stone D, Liraz-Zaltsman S, Mazzitelli J, Arenas M, Abduljawad N, Kliper E, Korczyn AD, Thareja NS, Kesner EL, Zhou M, Huang S, Silva TK, Katz N, Bornstein NM, Silva AJ, Shohami E, Carmichael ST. CCR5 Is a Therapeutic Target for Recovery after Stroke and Traumatic Brain Injury. Cell. 2019 Feb 21;176(5):1143-1157.e13. doi: 10.1016/j.cell.2019.01.044. PMID 30794775
- [Background] Lohse K, Bland MD, Lang CE. Quantifying Change During Outpatient Stroke Rehabilitation: A Retrospective Regression Analysis. Arch Phys Med Rehabil. 2016 Sep;97(9):1423-1430.e1. doi: 10.1016/j.apmr.2016.03.021. Epub 2016 Apr 22. PMID 27109329
- [Background] Zhou M, Greenhill S, Huang S, Silva TK, Sano Y, Wu S, Cai Y, Nagaoka Y, Sehgal M, Cai DJ, Lee YS, Fox K, Silva AJ. CCR5 is a suppressor for cortical plasticity and hippocampal learning and memory. Elife. 2016 Dec 20;5:e20985. doi: 10.7554/eLife.20985. PMID 27996938
- See also: Product Monograph for Celsentri (Maraviroc) — https://viivhealthcare.com/content/dam/cf-viiv/viiv-healthcare/en_CA/pdf/celsentri.pdf.pdf